CLINICAL TRIAL: NCT03099174
Title: An Open Label, Phase Ib, Dose-escalation Study Evaluating the Safety and Tolerability of Xentuzumab and Abemaciclib in Patients With Locally Advanced or Metastatic Solid Tumours and in Combination With Endocrine Therapy in Patients With Locally Advanced or Metastatic Hormone Receptor-positive, HER2-, Breast Cancer, Followed by Expansion Cohorts.
Brief Title: This Study in Patients With Different Types of Cancer (Solid Tumours) Aims to Find a Safe Dose of Xentuzumab in Combination With Abemaciclib With or Without Hormonal Therapies. The Study Also Tests How Effective These Medicines Are in Patients With Lung and Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1280.18; 2016-003142-85 (EudraCT Number)
Record Dates: First submitted 2017-03-31; First posted 2017-04-04 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Neoplasms; Breast Neoplasms
MeSH Terms: conditions — Neoplasms; Breast Neoplasms | interventions — xentuzumab; abemaciclib; Letrozole; Anastrozole; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort A: Xentuzumab 1000 mg & 150 mg Abemaciclib (Experimental): Patients with solid tumours received 1000 milligram (mg) Xentuzumab (weekly 10 mg/milliliter intravenous infusion) and 150 mg Abemaciclib (every 12 hours three 50 mg film coated tablets) in a 28-day cycle until disease progression, intolerability of the study medication, or consent withdrawal.
  Interventions: Drug: Xentuzumab; Drug: Abemaciclib
- Cohort B: Xentuzumab 1000 mg & 150 mg Abemaciclib & 2.5 mg Letrozole (Experimental): Patients with Hormone receptor+ (HR+) Human epidermal growth factor receptor 2 (HER2-) breast cancer received 1000 milligram (mg) Xentuzumab (weekly 10 mg/milliliter intravenous infusion) and 150 mg Abemaciclib (every 12 hours three 50 mg film coated tablets) in a 28-day cycle until disease progression, intolerability of the study medication, or consent withdrawal. Combined with a background therapy of 2.5 mg Letrozole (once daily film-coated tablet).
  Interventions: Drug: Xentuzumab; Drug: Abemaciclib; Drug: Letrozole
- Cohort C: Xentuzumab 1000 mg & 150 mg Abemaciclib & 1 mg Anastrozole (Experimental): Patients with Hormone receptor+ (HR+) Human epidermal growth factor receptor 2 (HER2-) breast cancer received 1000 milligram (mg) Xentuzumab (weekly 10 mg/milliliter intravenous infusion) and 150 mg Abemaciclib (every 12 hours three 50 mg film coated tablets) in a 28-day cycle until disease progression, intolerability of the study medication, or consent withdrawal. Combined with a background therapy of 1 mg Anastrozole (once daily film-coated tablet).
  Interventions: Drug: Xentuzumab; Drug: Abemaciclib; Drug: Anastrozole
- Cohort D: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant (Experimental): Patients with Hormone receptor+ (HR+) Human epidermal growth factor receptor 2 (HER2-) breast cancer received 1000 milligram (mg) Xentuzumab (weekly 10 mg/milliliter intravenous infusion) and 150 mg Abemaciclib (every 12 hours three 50 mg film coated tablets) in a 28-day cycle until disease progression, intolerability of the study medication, or consent withdrawal. Combined with a background therapy of 500 mg Fulvestrant (Faslodex®) (once a month intramuscular injection, with an additional 500 mg dose given two weeks after the first dose).
  Interventions: Drug: Xentuzumab; Drug: Abemaciclib; Drug: Fulvestrant
- Cohort E: Xentuzumab 1000 mg & 150 mg Abemaciclib (Experimental): Patients with non-small cell lung cancer (NSCLC) received 1000 milligram (mg) Xentuzumab (weekly 10 mg/milliliter intravenous infusion) and 150 mg Abemaciclib (every 12 hours three 50 mg film coated tablets) in a 28-day cycle until disease progression, intolerability of the study medication, or consent withdrawal.
  Interventions: Drug: Xentuzumab; Drug: Abemaciclib
- Cohort F: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant (Experimental): Patients with HR+ HER2- breast cancer & non-visceral disease received 1000 milligram (mg) Xentuzumab (weekly 10 mg/milliliter intravenous infusion) and 150 mg Abemaciclib (every 12 hours three 50 mg film coated tablets) in a 28-day cycle until disease progression, intolerability of the study medication, or consent withdrawal. Combined with a background therapy of 500 mg Fulvestrant (Faslodex®) (once a month intramuscular injection, with an additional 500 mg dose given two weeks after the first dose).
  Interventions: Drug: Xentuzumab; Drug: Fulvestrant; Drug: Abemaciclib
- Cohort D1: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant (Experimental): Patients with HR+ HER2- breast cancer & with visceral disease received 1000 milligram (mg) Xentuzumab (weekly 10 mg/milliliter intravenous infusion) and 150 mg Abemaciclib (every 12 hours three 50 mg film coated tablets) in a 28-day cycle until disease progression, intolerability of the study medication, or consent withdrawal. Combined with a background therapy of 500 mg Fulvestrant (Faslodex®) (once a month intramuscular injection, with an additional 500 mg dose given two weeks after the first dose).
  Interventions: Drug: Xentuzumab; Drug: Fulvestrant; Drug: Abemaciclib
- Cohort D2: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant (Experimental): Patients with HR+ HER2- breast cancer & with non-visceral disease received 1000 milligram (mg) Xentuzumab (weekly 10 mg/milliliter intravenous infusion) and 150 mg Abemaciclib (every 12 hours three 50 mg film coated tablets) in a 28-day cycle until disease progression, intolerability of the study medication, or consent withdrawal. Combined with a background therapy of 500 mg Fulvestrant (Faslodex®) (once a month intramuscular injection, with an additional 500 mg dose given two weeks after the first dose).
  Interventions: Drug: Xentuzumab; Drug: Fulvestrant; Drug: Abemaciclib

INTERVENTIONS:
Drug: Xentuzumab — Once weekly administrated through one hour intravenous infusion
Drug: Abemaciclib — Treatment/28-day cycle p.o. Q12H on Days 1-28 (dose determined in Cohort A) Abbreviations: PO = orally; Q12H = every 12 (± 2) hours
  Arms: Cohort A: Xentuzumab 1000 mg & 150 mg Abemaciclib; Cohort B: Xentuzumab 1000 mg & 150 mg Abemaciclib & 2.5 mg Letrozole; Cohort C: Xentuzumab 1000 mg & 150 mg Abemaciclib & 1 mg Anastrozole; Cohort D: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant; Cohort E: Xentuzumab 1000 mg & 150 mg Abemaciclib
Drug: Letrozole — Once a day
  Arms: Cohort B: Xentuzumab 1000 mg & 150 mg Abemaciclib & 2.5 mg Letrozole
Drug: Anastrozole — Once a day
  Arms: Cohort C: Xentuzumab 1000 mg & 150 mg Abemaciclib & 1 mg Anastrozole
Drug: Fulvestrant — Once a month, with an additional dose given two weeks after the first dose. Each dose is given as two slow injections lasting one to two minutes, with one injection being given into the muscle of each buttock
  Arms: Cohort D1: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant; Cohort D2: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant; Cohort D: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant; Cohort F: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant
Drug: Abemaciclib — Treatment/28-day cycle p.o. Q12H on Days 1-28 (dose determined in Cohort D) Abbreviations: PO = orally; Q12H = every 12 (± 2) hours
  Arms: Cohort D1: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant; Cohort D2: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant; Cohort F: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant

SUMMARY:
This is a study in adult patients with different types of cancer. The purpose of this study is to find a safe dose of:

* Xentuzumab in combination with abemaciclib
* Xentuzumab in combination with abemaciclib and hormonal therapies The study also tests whether these medicines make tumours shrink in participants with lung and breast cancer.

Participants can stay in the study as long as they benefit from and can tolerate treatment. All participants get xentuzumab infusions and abemaciclib tablets. Participants who have breast cancer get different types of hormonal therapies in addition to xentuzumab and abemaciclib.

For all participants, the size of the tumour is measured regularly. Doctors also regularly check the general health of the participants."

ELIGIBILITY:
Inclusion Criteria

All Cohorts

* Age ≥ 18 years (≥20 years for Japan only) at screening
* Signed and dated written informed consent in accordance with GCP (Good Clinical Practice ) and local legislation prior to admission to the trial
* WHO/ECOG (World Health Organization / Eastern Cooperative Oncology Group) performance status 0-1 assessed at screening
* Patient must be able to swallow oral capsules or tablets

Cohort A (Solid Tumours) & Cohort E (NSCLC):

- Male or female patients ready and able to use highly effective methods of birth control during the study and for 3 weeks following the last dose of abemaciclib per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information. Women of childbearing potential must have a negative serum pregnancy test at screening.

Cohort A (Solid Tumours)

* Patients with histologically or cytologically confirmed diagnosis of advanced and/or metastatic, measurable or evaluable, non-resectable solid tumours
* Patients must have received and failed, or have been intolerant to, all treatment known to confer clinical benefit or have no therapeutic options available as deemed appropriate by their treating physician
* Life expectancy ≥ 3 months in the opinion of the investigator assessed at screening;

Cohorts B, C, D (dose finding, Breast Cancer) & Cohort D1 and Cohort D2 (Breast Cancer):

* Women who have postmenopausal status due to either surgical/natural menopause or chemical ovarian suppression (initiated at least 28 days prior to Day 1 of Cycle 1) with a gonadotropin-releasing hormone (GnRH) agonist such as goserelin or radiation-induced ovarian suppression.

  -- postmenopausal status due to surgical/natural menopause requires at least one of the following conditions:
* prior bilateral oophorectomy
* age ≥ 60 years
* age < 60 years and amenorrheic (in the absence of tamoxifen, toremifene, ovarian suppression, or chemotherapy) for at least 12 months; and follicle-stimulating hormone (FSH) and estradiol within the postmenopausal range as per institutional reference ranges.
* Postmenopausal status due to radiation-induced ovarian suppression must be confirmed by FSH and estradiol level in the postmenopausal range.
* Histologically or cytologically proven diagnosis of breast cancer with evidence of locally advanced disease not amenable to curative resection or metastatic disease
* HR+ (local lab results at screening or, if not available, at the time of diagnosis) To fulfil the requirement of HR+ disease, the primary tumour or metastatic lesion of the breast cancer must express at least one of the hormone receptors (estrogen receptor [ER] or progesterone receptor [PgR]) by immunohistochemistry (IHC). Estrogen receptor and PgR assays are considered positive if there are at least 1% positive tumour nuclei in the sample as defined in the relevant American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) Guidelines (Hammond et al. 2010).
* HER2 negative (local lab results at screening or, if not available, at the time of diagnosis) as defined by the most recent American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) Guidelines (Hammond et al. 2010).

Cohorts B, C, D (dose finding), F (Breast Cancer):

* Previous adjuvant and neoadjuvant chemotherapy is permitted. 0-2 prior lines of chemotherapy for the metastatic setting are allowed (except Cohorts D1, D2 and F).
* At least 1 lesion (measurable or non-measurable) that can be accurately assessed at baseline with CT or MRI or PET-CT (CT portion of diagnostic quality) and which is suitable for accurate repeated measurement.
* Cohort B, C, D: Must be eligible for the corresponding hormonal therapy (letrozole, anastrozole or fulvestrant). For Cohorts B and C previous treatment with fulvestrant or exemestane is allowed. For For Cohort D, prior therapy with non steroidal aromatase inhibitors (anastrozole, letrozole) or exemestane are permitted.

Cohort E (NSCLC (Non-Small Cell Lung Cancer)):

* Histologically or cytologically confirmed diagnosis of stage IV NSCLC.
* The participant must have progressed after platinum-based chemotherapy AND immunotherapy (unless deemed inappropriate candidates for immunotherapy by their treating physician) AND have received 1 or a maximum of 2 other prior chemotherapy for advanced and/or metastatic disease OR must be judged by the physician as ineligible for further standard second-line chemotherapy. Prior treatment with epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI) and anaplastic lymphoma kinase (ALK) inhibitors is mandatory in participants whose tumour has EGFR-activating mutations or ALK translocations. Prior targeting agents and neoadjuvant/adjuvant therapies are permitted.
* Have adequate organ function including haematology, renal, and liver.
* Have measureable disease per RECIST 1.1.

Cohort D1, Cohort D2 and Cohort F (Breast Cancer):

* Have a negative serum pregnancy test at baseline (within 14 days prior to randomization) and agree to use medically approved precautions to prevent pregnancy during the study and for 3 weeks following the last dose of abemaciclib and for at least 6 months after last dose of xentuzumab if postmenopausal status is due to ovarian suppression with a GnRH agonist.
* Have either measurable disease or non-measurable bone only disease. Measurable and non-measurable diseases are defined according to the Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1 [v1.1]. Non-measurable bone only disease may include any of the following: blastic bone lesions, lytic bone lesions without a measurable soft tissue component, or mixed lytic-blastic bone lesions without a measurable soft tissue component.

Cohort D1 and D2 only:

* Patients must fulfil 1 of the following criteria:

  -- Relapsed with radiologic evidence of progression while receiving neoadjuvant or adjuvant endocrine therapy, with no subsequent endocrine therapy received following progression.
* Relapsed with radiologic evidence of progression within 1 year from completion of adjuvant endocrine therapy, with no subsequent endocrine therapy received following progression.
* Relapsed with radiologic evidence of progression more than 1 year from completion of adjuvant endocrine therapy and then subsequently relapsed with radiologic evidence of progression after receiving treatment with either an anti-estrogen or an aromatase inhibitor as first-line endocrine therapy for metastatic disease. Patients may not have received more than 1 line of endocrine therapy or any prior chemotherapy for metastatic disease.
* Presented de novo with metastatic disease and then relapsed with radiologic evidence of progression after receiving treatment with either an anti-estrogen or an aromatase inhibitor as first-line endocrine therapy for metastatic disease.

Patients may not have received more than 1 line of endocrine therapy or any prior chemotherapy for metastatic disease.

- For cohort D1 (visceral disease) patient must have at least one documented visceral metastasis; for cohort D2 (non-visceral disease), patient must not have any visceral metastasis.

Cohort F only:

* Patients with resistance to prior therapy with an aromatase inhibitor (AI) and CDK4/6 inhibitor (excluding abemaciclib) for locally advanced or metastatic breast cancer, defined as radiologic evidence of disease progression while on, or within 30 days after last dose of AI and/or CDK4/6 inhibitor (excl. abemaciclib) administered as first-line therapy for locally advanced or metastatic disease. Patients may not have received more than 1 line of prior endocrine based therapy or any prior chemotherapy for advanced/metastatic disease.
* Patient must not have any visceral metastasis (example of allowed lesions are in breast, lymph nodes, soft tissue, bone).

Exclusion criteria

All - Cohorts A, B, C, D (dose finding), E and F & Cohort D1 and Cohort D2 (Breast Cancer):

* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial
* Previous treatment in this trial
* Currently enrolled in another investigational device or drug study, or less than 21 days since ending another investigational device or drug study(s), or receiving other investigational treatment(s).
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable study subject or unlikely to complete the trial
* Prior anti-cancer chemotherapy, biological or radiation therapy, androgens, thalidomide, other anticancer agents, or any investigational drug within 21 days (14 days for non-myelosuppressive agents); and/or 4 weeks for immunotherapy, before starting any of the trial drugs.
* Prior radiotherapy to ≥ 25% of bone marrow regardless of when it was received
* Unresolved treatment related toxicity from previous therapy of > CTCAE grade 1 at study entry (except for stable sensory neuropathy ≤ CTCAE grade 2 and alopecia)
* Previous treatment with IGF-1R targeting compounds
* The patient has serious and/or uncontrolled pre-existing medical condition(s) that, in the judgement of the Investigator, would preclude participation in this study, including interstitial lung disease, severe dyspnoea at rest or requiring oxygen therapy.
* Inadequate bone marrow reserve or organ function as demonstrated by any of the following: ANC < 1.5 x 10^9/L, platelets < 100 x 10^9/L, haemoglobin <90g/L, ALT > 2.5 x ULN or > 5 x ULN in the presence of liver metastases, total bilirubin >1.5 x ULN or >3 x ULN in patients with Gilbert's syndrome, serum creatinine > 1.5 x ULN concurrent with creatinine clearance ≤ 50 mL/min.
* Pre-existing renal disease including glomerulonephritis, nephritic syndrome, Fanconi Syndrome or renal tubular acidosis
* Refractory nausea and vomiting, chronic GI diseases, inability to swallow the product, or previous significant bowel resection that would preclude adequate absorption of abemaciclib or resulting in baseline Grade 2 or higher diarrhoea
* Patients with Diabetes Type I or uncontrolled Type II (defined by HgBA1C > 8%).
* Patients with advanced/metastatic, symptomatic, visceral spread, that are at risk of life-threatening complications in the short term including patients with massive uncontrolled effusions (pleural, pericardial, peritoneal), pulmonary lymphangitis, and over 50% of liver involvement in metastases.
* Prior hematopoietic stem cell or bone marrow transplant
* Have a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia (including but not limited to ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest. Subjects with controlled atrial fibrillation for >30 days prior to study treatment are eligible.
* Erythropoietin, G-CSF, and GM-CSF are not allowed within 2 weeks prior to study. The primary prophylactic use of G-CSF is not permitted but it may be used to treat treatment emergent neutropenia.
* Have had major surgery (excluding biopsy) < 28 days of the initial dose of any of the study drugs or planned major surgery during study participation.
* Have active bacterial or fungal infection (that is, requiring IV antibiotics or therapy at time of initiating study treatment), and/or known viral infection (for example, human immunodeficiency virus [HIV] antibodies, hepatitis B surface antigen, or hepatitis C antibodies). Screening is not required for enrolment.
* Patients with baseline Grade ≥2 hyperglycaemia or patients with baseline Grade ≥ 2 diarrhoea
* Patients needing treatment with CYP3A4 inhibitors/inducers cannot be included in the trial.

Cohorts A, B, C, D (dose finding), E and F

* Any documented active or suspected malignancy or history of malignancy, other than the disease under study, within 3 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix or ductal carcinoma in situ (DCIS) if properly treated in opinion of the investigator.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial. Men who plan to father a child while in the trial.
* Prior anti CDK agents
* Known active uncontrolled or symptomatic CNS metastases, carcinomatous meningitis, or leptomeningeal disease, as indicated by clinical symptoms, cerebral oedema, and/or progressive growth. History of CNS metastases or cord compression are eligible if they have been definitively treated (e.g. radiotherapy, stereotactic surgery) and are clinically stable, off anticonvulsants and steroids for at least 4 weeks. Patients with brain metastases are eligible if they are asymptomatic, completed radiotherapy for at least 4 weeks or are on a stable dose of steroids for at least 4 weeks. Patients are not eligible if they have spinal cord compression.
* History of hypersensitivity to active or inactive excipients of xentuzumab, abemaciclib or letrozole/anastrozole/fulvestrant, or loperamide hydrochloride, or drugs with similar chemical structures

Cohort D1, Cohort D2 and Cohort F (Breast Cancer):

* Any documented active or suspected malignancy or history of malignancy (including inflammatory breast cancer), other than the disease under study, within 3 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix or ductal carcinoma in situ (DCIS) if properly treated in opinion of the investigator.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
* Have received prior treatment with chemotherapy (except for neoadjuvant/adjuvant chemotherapy), fulvestrant, everolimus, alpelisib or abemaciclib. For cohorts D1 and D2 only: prior treatment with palbociclib or ribociclib is also excluded)
* Have clinical evidence or history of central nervous system metastasis. Screening is not required for enrolment.
* History of hypersensitivity to active or inactive excipients of xentuzumab, abemaciclib or fulvestrant, or loperamide hydrochloride, or drugs with similar chemical structures
* Have initiated bisphosphonates or approved RANK ligand (RANK-L) targeted agents (for example, denosumab) <7 days prior to initiation of any study drug.
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (30):
- United States (6):
  - University of California Los Angeles, Santa Monica, California
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - University of Minnesota, Minneapolis, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
- Denmark (2):
  - Herlev and Gentofte Hospital, Herlev
  - Copenhagen University Hospital, Rigshospitalet, København Ø
- Finland (4):
  - Docrates Clinic, Helsinki
  - HUCH Comprehensive Cancer Center, building 2, Helsinki
  - Tampere University Hospital, Tampere
  - CRST - Clinical Research Services Turku, Turku
- France (4):
  - HOP Jean Minjoz, Besançon
  - INS Paoli-Calmettes, Marseille
  - INS Curie, Paris
  - Ctr Cario, Plerin Sur Mer
- Japan (4):
  - Aichi Cancer Center Hospital, Aichi, Nagoya
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - Tokai University Hospital, Kanagawa, Isehara
  - National Cancer Center Hospital, Tokyo, Chuo-ku
- South Korea (2):
  - National Cancer Center, Goyang
  - Severance Hospital, Seoul
- Spain (8):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Clínica Universidad de Navarra - Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Quirónsalud Madrid, Pozuelo de Alarcón

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website. The data shared are the raw clinical study data sets
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was an open label, phase Ib, dose-escalation study followed by expansion cohorts.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Cohort F: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant; Cohort D2: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant: Patients with non-visceral disease received 1000 milligram (mg) Xentuzumab (weekly 10 mg/milliliter intravenous infusion) and 150 mg Abemaciclib (every 12 hours three 50 mg film coated tablets) in a 28-day cycle until disease progression, intolerability of the study medication, or consent withdrawal. Combined with a background therapy of 500 mg Fulvestrant (Faslodex®) (once a month intramuscular injection, with an additional 500 mg dose given two weeks after the first dose).
- Cohort D1: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant: Patients with visceral disease received 1000 milligram (mg) Xentuzumab (weekly 10 mg/milliliter intravenous infusion) and 150 mg Abemaciclib (every 12 hours three 50 mg film coated tablets) in a 28-day cycle until disease progression, intolerability of the study medication, or consent withdrawal. Combined with a background therapy of 500 mg Fulvestrant (Faslodex®) (once a month intramuscular injection, with an additional 500 mg dose given two weeks after the first dose).
Period: Overall Study
Arm/Group | Cohort A: Xentuzumab 1000 mg & 150 mg Abemaciclib | Cohort B: Xentuzumab 1000 mg & 150 mg Abemaciclib & 2.5 mg Letrozole | Cohort C: Xentuzumab 1000 mg & 150 mg Abemaciclib & 1 mg Anastrozole | Cohort D: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort E: Xentuzumab 1000 mg & 150 mg Abemaciclib | Cohort F: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort D1: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort D2: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant
Started | 6 | 7 | 7 | 8 | 26 | 15 | 33 | 31
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 7 | 7 | 8 | 26 | 15 | 33 | 31
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 4
Not completed — Adverse Event | 0 | 1 | 1 | 2 | 5 | 3 | 6 | 4
Not completed — Other than listed | 6 | 6 | 5 | 6 | 19 | 10 | 26 | 23

BASELINE CHARACTERISTICS:
Population: Treated set (TS): all patients who are documented to have received and taken at least one dose of any study medication during the treatment cycles (including run-in period).
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Xentuzumab 1000 mg & 150 mg Abemaciclib | Cohort B: Xentuzumab 1000 mg & 150 mg Abemaciclib & 2.5 mg Letrozole | Cohort C: Xentuzumab 1000 mg & 150 mg Abemaciclib & 1 mg Anastrozole | Cohort D: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort E: Xentuzumab 1000 mg & 150 mg Abemaciclib | Cohort F: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort D1: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort D2: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Total
Number analyzed (Participants) | 6 | 7 | 7 | 8 | 26 | 15 | 33 | 31 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (3.6) | 53.6 (10.3) | 60.1 (12.5) | 51.9 (11.4) | 64.4 (7.0) | 56.7 (12.0) | 58.3 (10.2) | 53.7 (10.7) | 57.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 7 | 8 | 8 | 15 | 33 | 31 | 114
  Male | 1 | 0 | 0 | 0 | 18 | 0 | 0 | 0 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3
  Not Hispanic or Latino | 4 | 7 | 6 | 6 | 22 | 8 | 30 | 27 | 110
  Unknown or Not Reported | 2 | 0 | 1 | 2 | 3 | 6 | 3 | 3 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 2 | 4 | 1 | 9 | 7 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 2 | 5 | 5 | 4 | 17 | 8 | 21 | 21 | 83
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 1 | 2 | 4 | 6 | 3 | 3 | 22

OUTCOME MEASURES:

1. Primary Outcome: [Cohort A, B, C & D] Maximum Tolerated Dose (MTD) of Xentuzumab
Description: MTD during the MTD evaluation period (the first 28 day cycle). The MTD is defined as the highest dose with <25% risk of the true Dose limiting toxicity (DLT) rate >33%.
  DLT: adverse event or laboratory abnormality which 1) is related, probably related or possibly related to study drug and 2) meets any of the following criteria, unless that toxicity can be attributed to cancer progression or to identified etiology:
  CTCAE grade (Gr). 3+ hyperglycaemia (>48 hours), Gr. 4 hyperglycaemia, hematologic toxicity (>5 days), Gr. 3+ pneumonitis, febrile neutropenia, thrombocytopenia (Gr. 4 any duration, Gr. 3 w/ bleeding), AST/ALT > 5x ULN or > (baseline + 4x ULN), Gr. 3+ diarrhoea, nausea, vomiting (>2 days), skin rash, fatigue/asthenia (>7 days), Gr. 3-4 hyperlipidaemia (>2 weeks), Any AE causing 2-week treatment interruption, non-hematologic toxicities Gr. 3+ (except alopecia, infusion-related reaction), Any significant drug related toxicity qualified as DLT.
Time Frame: The first treatment cycle, up to 28 days.
Population: The MTD set defines the set of patients in the dose-finding cohorts (cohorts A,B,C and D) of the trial that are fully evaluable for determination of the MTD in the first treatment course.
Measure: Number; unit: milligram
Arm/Group | Cohort A: Xentuzumab 1000 mg & 150 mg Abemaciclib | Cohort B: Xentuzumab 1000 mg & 150 mg Abemaciclib & 2.5 mg Letrozole | Cohort C: Xentuzumab 1000 mg & 150 mg Abemaciclib & 1 mg Anastrozole | Cohort D: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant
Number analyzed (Participants) | 6 | 6 | 6 | 6
milligram | 1000 | 1000 | 1000 | 1000

2. Primary Outcome: [Cohort A, B, C & D] Number of Patients With DLTs in the MTD Evaluation Period
Description: Number of patients with Dose limiting toxicities in the MTD evaluation period.
  Dose limiting toxicity (DLT): adverse event or laboratory abnormality which 1) is related, probably related or possibly related to study drug and 2) meets any of the following criteria, unless that toxicity can be attributed to cancer progression or to identified etiology:
  CTCAE grade (Gr). 3+ hyperglycaemia (>48 hours), Gr. 4 hyperglycaemia, hematologic toxicity (>5 days), Gr. 3+ pneumonitis, febrile neutropenia, thrombocytopenia (Gr. 4 any duration, Gr. 3 w/ bleeding), AST/ALT > 5x ULN or > (baseline + 4x ULN), Gr. 3+ diarrhoea, nausea, vomiting (>2 days), skin rash, fatigue/asthenia (>7 days), Gr. 3-4 hyperlipidaemia (>2 weeks), Any AE causing 2-week treatment interruption, non-hematologic toxicities Gr. 3+ (except alopecia, infusion-related reaction), Any significant drug related toxicity qualified as DLT.
Time Frame: The first treatment cycle, up to 28 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Xentuzumab 1000 mg & 150 mg Abemaciclib | Cohort B: Xentuzumab 1000 mg & 150 mg Abemaciclib & 2.5 mg Letrozole | Cohort C: Xentuzumab 1000 mg & 150 mg Abemaciclib & 1 mg Anastrozole | Cohort D: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 2 | 1 | 1 | 1

3. Primary Outcome: [Cohort E] Number of Patients With Objective Response (OR)
Description: Objective response (OR) defined as best overall response of complete response (CR) or partial response (PR), where best overall response is determined according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 from date of first treatment administration (including run-in for cohort E) until the earliest of disease progression, death or last evaluable tumour assessment before start of subsequent anti-cancer therapy.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in short axis to <10 millimeter (mm)). For non-target lesions: disappearance of all non-target lesions and normalization of tumour marker level. All lymph nodes must be non-pathological in size (<10mm short axis).
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters.
Time Frame: Up to 26.5 months
Population: All patients in cohort E who were documented to have received and taken at least one dose of any study medication during the treatment cycles (including run-in period).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort E: Xentuzumab 1000 mg & 150 mg Abemaciclib
Number analyzed (Participants) | 26
Participants | 1

4. Primary Outcome: [Cohorts D1 and D2] Progression Free Survival (PFS) at 18 Months
Description: Progression free survival (PFS) rate at 18 month defined as the rate of absence of disease progression or death at the 18th month of treatment, where progression is determined according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1.
  Progression (PD): At least a 20% increase in the sum of diameters of target lesions, taking as references the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. For non-target lesions: Unequivocal progression of existing non-target lesions (Note: the appearance of one or more new lesions is also considered progression).
  Reported is the progression free survival rate at 18 months, based on a Kaplan-Meier.
Time Frame: Up to 18 months.
Population: All patients in cohort D1 and D2 who were documented to have received and taken at least one dose of any study medication during the treatment cycles (including run-in period).
Measure: Number; unit: Probability of Survival at 18 months
Arm/Group | Cohort D1: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort D2: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant
Number analyzed (Participants) | 33 | 31
Probability of Survival at 18 months | 0.4143 | 0.7854

5. Primary Outcome: [Cohort F] Disease Control (DC)
Description: Disease control (DC) defined as best overall response of complete response (CR) or partial response (PR) or confirmed stable disease (SD) (lasting for at least 24 weeks) or Non-CR/ Non-PD (lasting for at least 24 weeks) where best overall response is defined according to RECIST version 1.1 from first treatment administration until the earliest of disease progression, death or last evaluable tumour assessment before start of subsequent anti-cancer therapy.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as references the smallest sum diameters while on study.
Time Frame: Up to 18.5 months.
Population: All patients in cohort F who were documented to have received and taken at least one dose of any study medication during the treatment cycles (including run-in period).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort F: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant
Number analyzed (Participants) | 15
Participants | 6

6. Secondary Outcome: [Cohorts E, D1 and D2] Disease Control (DC)
Description: as for outcome 5
Time Frame: Up to 35.2 months.
Population: All patients in cohort Cohorts E, D1 and D2 who were documented to have received and taken at least one dose of any study medication during the treatment cycles (including run-in period).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort E: Xentuzumab 1000 mg & 150 mg Abemaciclib | Cohort D1: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort D2: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant
Number analyzed (Participants) | 26 | 33 | 31
Participants | 12 | 23 | 24

7. Secondary Outcome: [Cohorts E, F, D1 and D2] Time to Objective Response
Description: Time to objective response defined as the time from first treatment administration until first documented complete response (CR) or partial response (PR).
Time Frame: Up to 21.9 months.
Population: All patients in cohort Cohorts E, F, D1 and D2 who were documented to have received and taken at least one dose of any study medication during the treatment cycles (including run-in period) and who had an objective response.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cohort E: Xentuzumab 1000 mg & 150 mg Abemaciclib | Cohort F: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort D1: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort D2: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant
Number analyzed (Participants) | 1 | 1 | 20 | 6
Months | 1.94 [1.94 to 1.94] | 9.36 [9.36 to 9.36] | 3.52 [2.66 to 6.36] | 5.45 [1.71 to 14.23]

8. Secondary Outcome: [Cohorts E, F, D1 and D2] Duration of Objective Response
Description: Duration of objective response defined as the time from first documented complete response (CR) or partial response (PR) until the earliest of disease progression or death among patients with objective response.
Time Frame: Up to 27.2 months.
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cohort E: Xentuzumab 1000 mg & 150 mg Abemaciclib | Cohort F: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort D1: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort D2: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant
Number analyzed (Participants) | 1 | 1 | 20 | 6
Months | 5.78 [5.78 to 5.78] | 4.63 [4.63 to 4.63] | 11.12 [6.47 to 23.59] | 17.54 [11.17 to 23.95]

9. Secondary Outcome: [Cohorts E, F, D1 and D2] Duration of Disease Control
Description: Duration of disease control defined as the time from first treatment administration until the earliest of disease progression or death, among patients with disease control.
Time Frame: Up to 33.1 months.
Population: All patients in cohort Cohorts E, F, D1 and D2 who were documented to have received and taken at least one dose of any study medication during the treatment cycles (including run-in period) and who had disease control.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cohort E: Xentuzumab 1000 mg & 150 mg Abemaciclib | Cohort F: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort D1: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort D2: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant
Number analyzed (Participants) | 12 | 6 | 23 | 24
Months | 5.77 [2.68 to 6.85] | 12.42 [9.23 to 13.63] | 14.95 [10.87 to 24.67] | 22.01 [18.69 to 27.55]

10. Secondary Outcome: [Cohorts E, F, D1 and D2] Progression-free Survival (PFS)
Description: Progression-free survival (PFS) defined as the time from first treatment administration until tumour progression according to RECIST 1.1 or death from any cause, whichever occurs earlier.
  Progression (PD): At least a 20% increase in the sum of diameters of target lesions, taking as references the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. For non-target lesions: Unequivocal progression of existing non-target lesions (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 33 months.
Population: All patients in cohort Cohorts E, F, D1 and D2 who were documented to have received and taken at least one dose of any study medication during the treatment cycles (including run-in period).
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Cohort E: Xentuzumab 1000 mg & 150 mg Abemaciclib | Cohort F: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort D1: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort D2: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant
Number analyzed (Participants) | 26 | 15 | 33 | 31
Months | 2.1 [1.2 to 5.8] | NA [3.4 to NA] — Not enough patients with events. | 13.6 [4.5 to 30.2] | 33.1 [18.3 to 33.1]

11. Secondary Outcome: [Cohorts D1, D2 and F] Objective Response (OR)
Description: Objective response (OR) defined as best overall response of complete response (CR) or partial response (PR), where best overall response is determined according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 from date of first treatment administration until the earliest of disease progression, death or last evaluable tumour assessment before start of subsequent anti-cancer therapy.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in short axis to <10 millimeter (mm)). For non-target lesions: disappearance of all non-target lesions and normalization of tumour marker level. All lymph nodes must be non-pathological in size (<10mm short axis).
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters.
Time Frame: Up to 35.2 months.
Population: All patients in cohort Cohorts F, D1 and D2 who were documented to have received and taken at least one dose of any study medication during the treatment cycles (including run-in period).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort F: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort D1: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort D2: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant
Number analyzed (Participants) | 15 | 33 | 31
Participants | 1 | 20 | 6

ADVERSE EVENTS:
Time Frame: Up to approximately 35.5 months.
Description: Treated set (TS): all patients who were documented to have received and taken at least one dose of any study medication during the treatment cycles (including run-in period).
Arm/Group | Cohort A: Xentuzumab 1000 mg & 150 mg Abemaciclib | Cohort B: Xentuzumab 1000 mg & 150 mg Abemaciclib & 2.5 mg Letrozole | Cohort C: Xentuzumab 1000 mg & 150 mg Abemaciclib & 1 mg Anastrozole | Cohort D: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort E: Xentuzumab 1000 mg & 150 mg Abemaciclib | Cohort F: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort D1: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant | Cohort D2: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant
All-Cause Mortality (participants affected / at risk) | 2/6 | 2/7 | 2/7 | 0/8 | 13/26 | 1/15 | 5/33 | 1/31
Serious Adverse Events (participants affected / at risk) | 0/6 | 4/7 | 4/7 | 3/8 | 13/26 | 4/15 | 11/33 | 16/31
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 7/7 | 8/8 | 26/26 | 15/15 | 33/33 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Xentuzumab 1000 mg & 150 mg Abemaciclib (N=6) | Cohort B: Xentuzumab 1000 mg & 150 mg Abemaciclib & 2.5 mg Letrozole (N=7) | Cohort C: Xentuzumab 1000 mg & 150 mg Abemaciclib & 1 mg Anastrozole (N=7) | Cohort D: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant (N=8) | Cohort E: Xentuzumab 1000 mg & 150 mg Abemaciclib (N=26) | Cohort F: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant (N=15) | Cohort D1: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant (N=33) | Cohort D2: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant (N=31)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Implant site dehiscence (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis intestinal perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dry gangrene (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Xentuzumab 1000 mg & 150 mg Abemaciclib (N=6) | Cohort B: Xentuzumab 1000 mg & 150 mg Abemaciclib & 2.5 mg Letrozole (N=7) | Cohort C: Xentuzumab 1000 mg & 150 mg Abemaciclib & 1 mg Anastrozole (N=7) | Cohort D: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant (N=8) | Cohort E: Xentuzumab 1000 mg & 150 mg Abemaciclib (N=26) | Cohort F: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant (N=15) | Cohort D1: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant (N=33) | Cohort D2: Xentuzumab 1000 mg & 150 mg Abemaciclib & 500 mg Fulvestrant (N=31)
Anaemia (Blood and lymphatic system disorders) | 3 | 7 | 4 | 4 | 10 | 4 | 15 | 15
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 6 | 5 | 4 | 7 | 5 | 8 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 2 | 1 | 6 | 3 | 4 | 5
Bundle branch block left (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Conduction disorder (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 4
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 2
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 2
Eye haematoma (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 4
Photopsia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Xerophthalmia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 5 | 3 | 3 | 3 | 7 | 9 | 11
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3 | 3 | 1 | 0 | 0 | 6 | 6
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 2 | 3 | 2 | 10 | 9
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 7 | 6 | 8 | 16 | 14 | 30 | 29
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 5 | 5
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 4 | 3 | 1 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 4 | 4 | 6 | 16 | 4 | 22 | 21
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Retching (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 2 | 1 | 6 | 4
Teeth brittle (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 3
Vomiting (Gastrointestinal disorders) | 4 | 2 | 4 | 3 | 11 | 4 | 9 | 15
Asthenia (General disorders) | 3 | 5 | 5 | 5 | 6 | 9 | 12 | 10
Chest pain (General disorders) | 1 | 0 | 0 | 1 | 3 | 1 | 4 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2
Fatigue (General disorders) | 1 | 0 | 1 | 1 | 5 | 1 | 4 | 11
Feeling abnormal (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gait inability (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5
Injection site discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 3 | 1
Injection site pruritus (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 4
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 1
Nodule (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 5 | 2
Pain (General disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 2
Performance status decreased (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 2 | 2 | 2 | 5 | 6
Swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaccination site joint pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaccination site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Xerosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 5
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 3
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Dermatophytosis of nail (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 4
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 4 | 0 | 1 | 2 | 2
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1 | 1 | 1 | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 2 | 1 | 3 | 6 | 6
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Urostomy complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 4 | 1 | 0 | 3 | 2 | 7 | 7
Aspartate aminotransferase increased (Investigations) | 2 | 6 | 1 | 0 | 4 | 4 | 8 | 7
Basophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 4 | 1 | 0 | 0 | 1 | 3 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 3
Blood creatine phosphokinase MB increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 2 | 4 | 4
Blood creatinine increased (Investigations) | 2 | 3 | 4 | 3 | 8 | 2 | 8 | 8
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Blood urea increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram PR shortened (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 4 | 1 | 1 | 0 | 2 | 7 | 3
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Glomerular filtration rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 2 | 1 | 1 | 1 | 3 | 0 | 5 | 2
Neutrophil count decreased (Investigations) | 2 | 1 | 2 | 1 | 4 | 1 | 17 | 16
Platelet count decreased (Investigations) | 2 | 3 | 1 | 2 | 9 | 2 | 10 | 13
Protein total decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Weight decreased (Investigations) | 1 | 1 | 0 | 1 | 4 | 1 | 2 | 6
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
White blood cell count decreased (Investigations) | 2 | 2 | 1 | 1 | 8 | 0 | 8 | 7
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3 | 4 | 3 | 11 | 7 | 12 | 10
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 5 | 0 | 1 | 2
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 5
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 3 | 1 | 2 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 4 | 2 | 3 | 3 | 8 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 6 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 3 | 1 | 4 | 12 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 1 | 1 | 3 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 3 | 8 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3 | 1 | 4 | 4 | 5
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0 | 1 | 2 | 8 | 7
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 6 | 1
Headache (Nervous system disorders) | 1 | 2 | 1 | 3 | 0 | 8 | 12 | 15
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Occipital neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 2 | 1
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0
Apathy (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Depression (Psychiatric disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 3 | 1
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyssomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 1 | 0 | 2 | 6 | 7
Mood swings (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bladder pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 4 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 2
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 4 | 2 | 2 | 7 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 3 | 0 | 3 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 1 | 1 | 4 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 2 | 0 | 3 | 5
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 1
Erythrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Melanoderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 4 | 2
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1 | 2 | 2 | 8 | 5
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3 | 4 | 3 | 3 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4
Axillary vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 4 | 3
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 3 | 2
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT03099174/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT03099174/SAP_001.pdf